CLINICAL TRIAL: NCT07026955
Title: Colorectal Cancer in Young Adults: Study of Incidence, Survival, and Prognostic Factors in Tarragona, Spain
Acronym: CCR50
Status: Completed | Type: Observational
Sponsor: HJ23 (Industry)
Collaborators: Joan XXIII University Hospital (Other)
Responsible Party: Principal Investigator, Jordi Elvira Lopez, Principal investigator, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: CGD-HJ23; 009/2024 (Other: CEIm)
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer in Patients Under 50 Years of Age; Colorectal Cancer
Keywords: Colorectal cancer; cancer screening; early onset cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- colorectal cancer in patients under 50 years of age
  Interventions: Other: colorectal cancer in patients over 50 years of age

INTERVENTIONS:
Other: colorectal cancer in patients over 50 years of age — description

SUMMARY:
We conducted an observational, descriptive, longitudinal and retrospective study of 59 patients under 50 years of age diagnosed with CRC in the province of Tarragona, between 2019 and 2024. Sociodemographic, clinical, anatomopathological and evolutionary variables provided from the data collected in the registry of the Colorectal Cancer Committee of the Joan XXIII University Hospital (HJ23) were analyzed.

DETAILED DESCRIPTION:
Study Design

This descriptive, longitudinal, observational, retrospective study included patients under 50 diagnosed with colorectal cancer at HJ23 between 2019 and 2024. The protocol was approved by the CEIm IISPV (ref. 009/2024)

Study Population

Participants Data were obtained from patients under 50 years of age diagnosed with CRC and evaluated by the colorectal cancer multidisciplinary team (MDT) at the HJ23 during the period 2019-2024.

Inclusion criteria included all patients under 50 years of age diagnosed with CRC and evaluated by the MDT during the specified period.

Exclusion criteria comprised patients over 50 years of age, those with primary tumors of non-colorectal origin, and individuals diagnosed with polyps with low-grade dysplasia, hyperplastic polyps, or other non-neoplastic colorectal conditions.

Study Methods

Data were obtained from the registry of patients presented at the Multidisciplinary Colorectal Cancer Committee of the HJ23 between 2019 and 2024.

The hospital informatic team provided a refined list of medical record numbers for patients under 50 years of age evaluated by the committee.

The information was encoded into a password-protected Microsoft Access database hosted on the hospital intranet. Subsequently, detailed review of medical records was conducted, resulting in a pseudonymized dataset for analysis.

Study Variables Sociodemographic variables included sex (male or female), age (under 50), and referring hospital to assess the demographic distribution by origin.

Clinical characteristics included date of first symptom, reason for consultation, poor prognostic factors, and tumor staging using the TNM classification , based on clinical, imaging, and/or pathological data.

Management and follow-up variables included date of presentation to the MDT, the treatment decision taken, presence of local recurrence or metastases, date of last surgical follow-up, and, if applicable, date of death.

Diagnostic procedures included colonoscopy, date, distance from anal verge in centimeters, and histopathological findings. Imaging studies included the performance of CT scans, recording whether performed and the date of examination.

Surgical treatment variables included whether surgery was performed, date of surgery, surgical approach (open, laparoscopic, robotic).

Histopathological variables for operated patients included the pathological evaluation of the surgical specimen, TNM staging, lymphovascular invasion, distant metastases, tumor budding grade (low, intermediate, high, or not assessable), and MSH2/MSH6 mismatch repair protein expression (preserved/not preserved). Postoperative complications were classified using the Clavien-Dindo scale. Data on genetic counseling were also recorded, including conclusions on pathogenic variants, variants of uncertain significance, or benign findings.

Statistical Analysis Quantitative variables with a normal distribution were expressed as mean and standard deviation (SD); otherwise, they were presented as median and interquartile range (IQR). Categorical variables were described using mode and proportions. The Shapiro-Wilk test was used to assess the normality of continuous variables. A p-value < 0.05 was considered statistically significant. If normality was not confirmed, p-values were obtained using permutation tests.

Group comparisons were made using Fisher's exact test for categorical variables, and the Student's t-test or ANOVA for normally distributed quantitative variables. For non-normal distributions, the Wilcoxon-Mann-Whitney test was used for two groups, and the Kruskal-Wallis test for more than two groups. Fisher's and McNemar's tests were used for contingency tables, as appropriate.

All analyses were performed using STATA© (StataCorp), conducted by a statistician specialized in data processing and analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients under 50 years of age
* diagnosed: colorectal cancer

Exclusion Criteria:

* over 50 years of age,
* Primary tumors of non-colorectal origin
* individuals diagnosed with polyps with low-grade dysplasia, hyperplastic polyps
* other non-neoplastic colorectal conditions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all patients under 50 years of age diagnosed with colorectal cance
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
INCIDENCE | 5 year
  describe the incidence of colorectal cancer in individuals under 50 years of age in the population of the province of Tarragona.

SECONDARY OUTCOMES:
mortality | 5 years
  describe the mortality of colorectal cancer in individuals under 50 years of age in the population of the province of Tarragona.
survival | 5 years
  describe the survival of colorectal cancer in individuals under 50 years of age in the population of the province of Tarragona.
prognostic factor | 5 year
  describe the prognostic factor of colorectal cancer in individuals under 50 years of age in the population of the province of Tarragona.
cancer treatment | 5 year
  to describe the various medical and surgical treatments received by the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Tarragona Joan XXIII, Tarragona, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Yes
there ara a anonymous data, so we can share
Supporting Information: SAP
Time Frame: 1 year
Access Criteria: same study